CLINICAL TRIAL: NCT05178121
Title: Formative Evaluation of an eLearning Approach to Suicide Prevention Training
Brief Title: eLearning for Suicide Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Doyanne Darnell, Assistant Professor, School of Medicine: Psychiatry, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00013577; K23MH118361-01A1 (NIH)
Record Dates: First submitted 2021-10-08; First posted 2022-01-05 (Actual); Results first posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-11

CONDITIONS: Suicide
Keywords: Education; Suicide Prevention; Fidelity; Artificial Intelligence
MeSH Terms: conditions — Suicide; Suicide Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Project WISE eLearning Training in Suicide Safety Planning (Experimental)
  Interventions: Behavioral: eLearning Training in Suicide Safety Planning

INTERVENTIONS:
Behavioral: eLearning Training in Suicide Safety Planning — The training includes a web-based didactic in suicide safety planning, interactive practice in counseling microskills with a chat bot, role-playing safety planning with a standardized patient, and reviewing automated feedback on safety planning counseling skills generated from a computer coding system.

SUMMARY:
Project WISE (Workplace Integrated Support & Education) includes developmental and pilot research to create an e-learning training in suicide safety planning enhanced with novel skill-building technologies that can be integrated into the routine workflow of nurses serving patients hospitalized for medical, surgical, or traumatic injury reasons. This study pilots an initial version of this eLearning training and collects data on the acceptability of the training and its components as well as engagement of nurses in the training. The evaluation will inform iterations of the training.

ELIGIBILITY:
Inclusion Criteria:

* Nurses working in acute or intensive care units at Harborview Medical Center

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doyanne A Darnell, PhD, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Reporter — https://reporter.nih.gov/project-details/10210226

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Nurses recruited from medical center via email, flyer, and unit manager notifications of the study.
  Recruitment period: November 1, 2021 - May 31, 2022
Period: Overall Study
Arm/Group | Project WISE eLearning Training in Suicide Safety Planning
Started | 18 (Although 19 participants consented to participate in the study, one participant did not continue with participation after the consent and enrollment process.)
Completed Training | 15
Completed Post-Training Survey | 14
Completed Post-Training Role-Play | 14
Completed 6-Month Role-Play | 10
Completed (Completed 6-Month Follow-up Survey) | 13
Not Completed | 5
Not completed — Other | 4
Not completed — Data collection ended before participant reached 6 months | 1

BASELINE CHARACTERISTICS:
Population: 18 of 19 enrolled participants actually participated in the study and completed a baseline measure of demographics.
Arm/Group | Project WISE eLearning Training in Suicide Safety Planning
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Training Acceptability - System Usability Scale for Client Bot Emily
Description: The System Usability Scale, a self-report measure using a Likert-type rating scale, will assess acceptability of the two technologic training components: Client Bot Emily and Lyssn Advisor. Client Bot Emily is a virtual patient/chat bot with the persona of a suicidal patient. Nurses chat with Emily and practice skills of asking open-ended questions and making reflections about statements Emily makes. Lyssn Advisor is an online platform that automatically codes transcripts of audio or video recorded role-plays for counseling skills; nurses then log in to the platform to see their scores, which provides feedback on their counseling performance.
  Scores on the SUS range from 0-100, which higher scores indicating greater usability or acceptability.
Time Frame: Once, immediately after engaging with each of the training technologies
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Project WISE eLearning Training in Suicide Safety Planning: eLearning Training in Suicide Safety Planning: The training includes a web-based didactic in suicide safety planning, interactive practice in counseling microskills with a chat bot "Client Bot Emily", role-playing safety planning with a standardized patient, and reviewing automated feedback on safety planning counseling skills generated from a computer coding system (Lyssn Advisor).
Arm/Group | Project WISE eLearning Training in Suicide Safety Planning
Number analyzed (Participants) | 16
score on a scale | 70.3 (19.7)

2. Primary Outcome: Training Acceptability Self-Report - Post-Training
Description: A 4-item self-report measure created for this study will assess satisfaction with all of the training components using a Likert-type scale of 0 = Not at all satisfied to 4 = Completely satisfied.
Time Frame: Immediately after completing the training
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Project WISE eLearning Training in Suicide Safety Planning
Number analyzed (Participants) | 14
score on a scale
  Satisfaction with the didactic and demonstration | 3.1 (0.8)
  Satisfaction with Client Bot Emily | 1.1 (1.1)
  Satisfaction with the role-play practice | 3.5 (0.5)
  Satisfaction with the Lyssn Advisor feedback | 2.5 (0.6)

3. Primary Outcome: Training Acceptability Self-Report - 6-Month Follow-up
Description: as for outcome 2
Time Frame: 6-months after completing the training
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Project WISE eLearning Training in Suicide Safety Planning
Number analyzed (Participants) | 13
score on a scale
  Satisfaction with the didactic and demonstration | 3.2 (0.8)
  Satisfaction with Client Bot Emily | 1.5 (1.2)
  Satisfaction with the role-play practice | 3.5 (0.5)
  Satisfaction with the Lyssn Advisor feedback | 2.6 (1.0)

4. Primary Outcome: Training Engagement With Client Bot User Data - Post-Training
Description: Data is collected from the technologic platform on whether and how often participants accessed the training technologies. Engagement is indicated by participants accessing the platform using their unique login and interacting with the webpage associated with the Client Bot. The unit of measurement will be the number of participants who accessed the Client Bot during the training period.
Time Frame: Immediately after participants indicate they have completing the training activities
Measure: Count of Participants; unit: Participants
Arm/Group | Project WISE eLearning Training in Suicide Safety Planning
Number analyzed (Participants) | 18
Participants | 16

5. Primary Outcome: Training Engagement With Lyssn Advisor User Data - Post-Training
Description: Data is collected from the technologic platform on whether and how often participants accessed the training technologies. Engagement is indicated by participants accessing the platform using their unique login and interacting with the webpage associated with the Lyssn Advisor. The unit of measurement will be the frequency of times participants visits the Lyssn Advisor webpage.
Time Frame: Immediately after participants indicate they have completing the training activities
Population: We were unable to collect this data
Arm/Group | Project WISE eLearning Training in Suicide Safety Planning
Number analyzed (Participants) | 0

6. Primary Outcome: Training Engagement With Client Bot User Data - 6-Month Follow-up
Description: Data is collected from the technologic platform on whether and how often participants accessed the training technologies. Engagement is indicated by participants accessing the platform using their unique login and interacting with the webpage associated with the Client Bot. The unit of measurement will be the number of participants who logged on and interacted with the Client Bot after the training period and before completing the 6-month survey.
Time Frame: 6-months after participants indicate they have completed the training activities
Population: 16 participants interacted with Client Bot Emily during the training period.
Measure: Count of Participants; unit: Participants
Arm/Group | Project WISE eLearning Training in Suicide Safety Planning
Number analyzed (Participants) | 16
Participants | 0

7. Primary Outcome: Training Engagement With Lyssn Advisor User Data - 6-Month Follow-up
Description: Data is collected from the technologic platform on whether and how often participants accessed the training technologies. Engagement is indicated by participants accessing the platform using their unique login and interacting with the webpage associated with the Lyssn Advisor. The unit of measurement will be the frequency of times participants visits the Lyssn Advisor webpage during the 6-month follow-up period.
Time Frame: 6-months after participants indicate they have completed the training activities
Population: Participant login to the Lyssn system after initial training was not able to be captured, therefore, the outcome data for this variable were not collected.
Arm/Group | Project WISE eLearning Training in Suicide Safety Planning
Number analyzed (Participants) | 0

8. Primary Outcome: Training Engagement Self-Report - Post-Training
Description: Investigators will collect self-reported completion of the training activities using a 4-item measure. Participants will report on a sliding scale from 0-100, what percent of each training activity they believe they completed.
Time Frame: Immediately after participants indicate they have completed the training activities
Measure: Mean (Standard Deviation); unit: percentage of completion
Arm/Group | Project WISE eLearning Training in Suicide Safety Planning
Number analyzed (Participants) | 14
percentage of completion
  Percent completion of didactic and demonstration | 94.3 (14.4)
  Percent completion of Client Bot Emily activity | 81.8 (18.1)
  Percent completion of role-play practice | 95.3 (11.0)
  Percent completion of Lyssn Advisor activity | 90.5 (12.2)

9. Primary Outcome: Client Bot Training Engagement Self-Report - 6 Month Follow-up
Description: Participants will self-report whether or not they accessed any of the training technologies during the follow-up period.
Time Frame: 6-months after participants indicate they have completed the training activities
Measure: Count of Participants; unit: Participants
Arm/Group | Project WISE eLearning Training in Suicide Safety Planning
Number analyzed (Participants) | 13
Participants | 3

10. Primary Outcome: Participant Retention
Description: Percent of participants retained throughout study follow-up
Time Frame: 6 Months after completing the training
Population: 19 participants enrolled in the study; however, of these, 18 participants participated in some aspect of the study, including completed the baseline survey
Measure: Count of Participants; unit: Participants
Arm/Group | Project WISE eLearning Training in Suicide Safety Planning
Number analyzed (Participants) | 18
Participants
  Retained through the 6-month survey | 13
  Retained through the 6-month role-play | 10

11. Primary Outcome: Training Acceptability - System Usability Scale for Lyssn Advisor
Description: as for outcome 1
Time Frame: Once, immediately after engaging with each of the training technologies
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Project WISE eLearning Training in Suicide Safety Planning
Number analyzed (Participants) | 14
score on a scale | 65.4 (16.3)

12. Primary Outcome: Lyssn Advisor Training Engagement Self-Report - 6 Month Follow-up
Description: Participants will self-report whether or not they accessed any of the training technologies during the follow-up period.
Time Frame: 6-months after participants indicate they have completed the training activities
Population: 13 nurses completed the 6-month follow-up survey and therefore reported on technology use during that period of time.
Measure: Count of Participants; unit: Participants
Arm/Group | Project WISE eLearning Training in Suicide Safety Planning
Number analyzed (Participants) | 13
Participants | 6

ADVERSE EVENTS:
Time Frame: The time frame for participants in the study was expected to be 7 months from the baseline/pre-training survey to the 6-month post-training survey (1 month to complete the training activities).
Arm/Group | Project WISE eLearning Training in Suicide Safety Planning
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-09-17): https://cdn.clinicaltrials.gov/large-docs/21/NCT05178121/Prot_SAP_ICF_000.pdf